CLINICAL TRIAL: NCT03139812
Title: Effects of Daily Irrigation on Corneal Epithelial Permeability and Adverse Events With Silicone Hydrogel Contact Lens Continuous Wear
Brief Title: Daily Irrigation With Silicone Hydrogel Contact Lens Continuous Wear
Acronym: EW23
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: University of California, Berkeley (Other)
Responsible Party: Principal Investigator, Meng C. Lin, Associate Professor, Clinical Optometry and Vision Science Program, University of California, Berkeley
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: UCBCRCEW23
Record Dates: First submitted 2017-04-17; First posted 2017-05-04 (Actual); Last update posted 2017-05-04 (Actual); Status verified 2017-05

CONDITIONS: Corneal Epithelial Permeability
Keywords: continuous contact lens wear; silicone hydrogel contact lenses; irrigation; corneal epithelial permeability; contact lens-related adverse events

STUDY DESIGN:
Intervention Model Description: 161 non-contact lens wearers were fit with silicone hydrogel (SiH) contact lenses and randomized to either a treatment (n = 81) or control (n = 80) group for 30-day continuous wear (CW). Subjects in the treatment group irrigated every morning and whenever dryness symptoms occurred; subjects in the control group did not.
Who Masked: Investigator
Masking Description: Research optometrists conducting eye examinations and technicians conducting fluorometry measurements did not know whether a given subject was in the treatment (irrigating) or control (non-irrigating) group.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- 30-day SiH CW, No Daily Irrigation (Other): Control group subjects wore SiH lenses for 30-day CW under normal clinical practice guidelines with no daily morning irrigation of the eyes with sterile saline solution
  Interventions: Device: 30-day SiH CW
- 30-day SiH CW, Daily Irrigation (Other): Treatment group subjects wore SiH lenses for 30-day CW under normal clinical practice guidelines, and also irrigated the eyes with sterile saline solution every morning upon awakening
  Interventions: Drug: Daily irrigation; Device: 30-day SiH CW

INTERVENTIONS:
Drug: Daily irrigation — Daily morning irrigation of the eye with sterile, borate-buffered, saline solution (Unisol 4) and gentle nudging of the lens to promote solution flow beneath the lens
  Other Names: Unisol 4 (Alcon Laboratories, Inc., Fort Worth, TX)
  Arms: 30-day SiH CW, Daily Irrigation
Device: 30-day SiH CW — 30-day continuous wear of silicone hydrogel contact lenses

SUMMARY:
This study sought to determine whether daily irrigation with sterile saline solution during silicone hydrogel (SiH) contact lens continuous wear (CW) could improve ocular surface integrity and reduce the risk of adverse events.

DETAILED DESCRIPTION:
The purpose of this study was to determine whether daily irrigation with sterile saline solution during silicone hydrogel (SiH) contact lens 30-day continuous wear (CW) can mitigate increases in corneal epithelial permeability (Pdc) and reduce the risk of mechanical, contact lens-induced, inflammatory, and overall adverse events. 161 non-contact lens wearers were fit with SiH contact lenses and randomized to either a treatment (n = 81) or control (n = 80) group for 30-day CW. Subjects in the treatment group irrigated every morning and whenever dryness symptoms occurred; subjects in the control group did not.

ELIGIBILITY:
Inclusion Criteria:

* spectacle prescriptions between -1.00 diopter sphere (DS) and -10.00 DS;
* less than 0.75 diopters (D) of astigmatism;
* free of any ocular disease or systemic disease with ocular manifestation;

Exclusion Criteria:

* history of contact lens wear within the past year;
* history of ocular surgery or serious injury;
* presence of corneal scarring;
* frequent swimming, smoking, or use of medications w/ ocular side effects;

Ages: 18 Years to 39 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 161 (Actual)
Dates: Start 2012-01-15 (Actual); Primary Completion 2012-10-15 (Actual); Study Completion 2012-10-15 (Actual)

PRIMARY OUTCOMES:
Corneal epithelial permeability (Pdc) at Baseline | Baseline
  Rate of fluorescein clearance through the corneal epithelium, measured by scanning fluorometry, in nm/sec at baseline with no contact lenses
Corneal epithelial permeability (Pdc) Post-1-Day CW | Post-1-Day CW of SiH contact lenses
  Rate of fluorescein clearance through the corneal epithelium, measured by scanning fluorometry, in nm/sec after 1 night of contact lens CW
Corneal epithelial permeability (Pdc) Post-30-Day CW | Post-30-Day CW of SiH contact lenses
  Rate of fluorescein clearance through the corneal epithelium, measured by scanning fluorometry, in nm/sec after 30 nights of contact lens CW
Risk of adverse events | Post-30-day CW of SiH contact lenses
  Odds ratios (OR) for adverse events: contact lens-induced, mechanically-induced, inflammatory, and overall

CONTACTS AND LOCATIONS:
Overall Officials: Meng C Lin, OD, PhD, FAAO, Principal Investigator — University of California, Berkeley

REFERENCES:
- [Background] Lin MC, French HM, Graham AD, Sanders TL. Effects of daily irrigation on corneal epithelial permeability and adverse events with silicone hydrogel contact lens continuous wear. Invest Ophthalmol Vis Sci. 2014 Feb 10;55(2):776-83. doi: 10.1167/iovs.13-13508. PMID 24425854